CLINICAL TRIAL: NCT05600361
Title: 13C-Pyruvate DNP MR Spectroscopy for Detecting Early Treatment Response in Patients With Lymphoma
Brief Title: 13C Pyruvate DNP MR Spectroscopy for Lymphoma Treatment Response Assessment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOST 111-2314-B-182A-042
Record Dates: First submitted 2022-10-11; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Patient Outcome Assessment
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Using 13C pyruvate DNP MR spectroscopy to evaluate for early treatment response in patients with lymphoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients having 13C Pyruvate DNP for lymphoma early treatment response evaluate (Other): In stage 1, we expected to enroll 8 first-time diagnosed lymphoma patients referred from clinicians for 13C-pyruvate DNP MRS. In stage 2, another 8 patients with proven relapse will be referred from clinicians for 13C-pyruvate DNP MRS. We will collect related clinical information, patient follow up information, including treatment outcome, and imaging parameters from MRI and PET/CT.
  Interventions: Drug: hyperpolarized 13C-labeled pyruvate from dynamic nuclear polarization (DNP) magnetic resonance spectroscopy

INTERVENTIONS:
Drug: hyperpolarized 13C-labeled pyruvate from dynamic nuclear polarization (DNP) magnetic resonance spectroscopy — In stage 1, we expected to enroll 8 first-time diagnosed lymphoma patients referred from clinicians for 13C-pyruvate DNP MRS. In stage 2, another 8 patients with proven relapse will be referred from clinicians for 13C-pyruvate DNP MRS. We will collect related clinical information, patient follow up information, including treatment outcome, and imaging parameters from MRI and PET/CT.

SUMMARY:
This study has two stages and the aims are as follows:

Aim 1:

In Stage 1 of this study, the investigators aim to recruit first-time diagnosed lymphoma patients, to understand the changes of metabolites before and after treatment, and to evaluate the ability of hyperpolarized 13C-labeled pyruvate from dynamic nuclear polarization (DNP) magnetic resonance spectroscopy (MRS) for detecting early treatment response in these patients.

The pre-treatment metabolic imaging biomarker levels will be compared to the followings:

1. Post-treatment metabolites from 13C-pyruvate DNP MRS after the first week of chemotherapy
2. Interval change in tumor size
3. ADC values from diffusion weighted imaging (DWI), SUV values from 18F-FDG PET/CT before and after the first week of chemotherapy
4. Pre-treatment and interim follow up SUV values from 18F-FDG PET/CT
5. Post-treatment outcome and to understand the change of metabolites before and after treatment and if possible, evaluate treatment outcome using the above imaging biomarkers

Aim 2:

In Stage 2 of this study, the investigators aim to recruit lymphoma patients with proven relapse after treatment, to understand the changes of metabolites before and after treatment, to compare the metabolite changes with Stage 1 patients and to evaluate the ability of hyperpolarized 13C-labeled pyruvate from DNP MRS for detecting early treatment response in these patients.

DETAILED DESCRIPTION:
Background Information

Metabolites from aberrant metabolic pathways in lymphoma Cells can be detectable through DNP 13C Pyruvate MR Spectroscopy and its potential benefit in lymphoma patients

Lymphoma is a common cause of malignancy. The assessment of tumor response after treatment largely depends on comparison of the pre-treatment and post-treatment changes in tumor size, while more advanced imaging methods, such as metabolic imaging, are taking more important roles in early detection of tumor response. Moreover, early tumor response to treatment were also indicators of future clinical outcome. Measurement of changes in tumor size may be a non-invasive and simple method of evaluating treatment response, but this method lacks sensitivity because some patients may require more than several weeks before evidence of tumor shrinkage can be shown. In addition, tumor treatment may result in a stasis of tumor size, which the differentiation between post-treatment residual tumor from non-viable mass may also be challenging. If the tumor is not responding, a more effective treatment regimen could be initiated; rapidly changing the patient to a more effective drug not only is cost-effective but also can greatly improve morbidity and mortality.

Metabolic imaging of tumor utilizes the metabolic dominance of tumor through the glycolysis process, which is the Warburg effect. Similar to 18F-FDG PET/CT, which glycolysis is upregulated between in malignant tumor as compared to normal tissue; Pyruvate, the intermediate metabolite from glycolysis and the main substrate for our study, can be further metabolized according to the pathways:

(A) Lactate through the lactate dehydrogenate pathway which is the main target for the analysis in our study (B) Bicarbonate (HCO3) through the nicotinamide adenine dinucleotide (NAD) <--> NADH (H for hydrogen) pathway (C) Glutamate and Alanine through the tricarboxylic acid cycle (TCA) cycle

The metabolic pathways described above are not one-way road, but rather the generation of metabolic intermediates can be conversed back and forth through enzymes, the metabolic pathways may be aberrant, and the flux of metabolites may be altered or upregulated by changes in cell environment and especially in the presence of tumor. The aberrant metabolism through aerobic glycolysis displayed by tumor cells provides opportunities for tumor detection and treatment response monitoring using metabolic imaging. Rather than downwards to the TCA cycle as normal cells would, cancer cells tend to upregulate the metabolism of pyruvate toward lactate production.

The changes in metabolite after glycolysis shown above is the foundation for development of advanced metabolic imaging in lymphoma; in which lymphoma cells were shown to upregulate the LDH-catalyzed interconversion from pyruvate to lactate. MRS is an ideal tool for the non-invasive study of metabolism due to the extensive range of compounds it can detect. 13C MRS, which can detect signals from multiple cellular metabolites following administration of a 13C-labelled substance, such as pyruvate, has been used to follow metabolic processes in vivo. Following the first pre-clinical study using DNP MRS of 13C-labeled substrate to increase their sensitivity of detection by >10,000 times, DNP MRS of 13C-pyruvate remains the main substrate for both pre-clinical animal studies and the recent human studies from cancers in various organs, such as the brain, kidney and prostate. These studies showed that despite no currently available clinical human research has been done in lymphoma patients using 13C-Pyruvate DNP MRS, this method is feasible in assessment of tumor treatment response from the lactate-to-pyruvate ratio in related pre-clinical animal lymphoma studies, with safety established in other clinical human studies.

Material and Methods

Patient enrollment and clinical data collection This study is to be performed in two stages and is expected to be completed in two years. In stage 1, the investigators expected to enroll 8 first-time diagnosed lymphoma patients referred from clinicians for 13C-pyruvate DNP MRS. In stage 2, another 8 patients with proven relapse will be referred from clinicians for 13C-pyruvate DNP MRS. The investigators will collect related clinical information, patient follow up information, including treatment outcome, and imaging parameters from MRI and PET/CT.

The patient enrollment inclusion criteria include:

1. Able to understand and provide signed informed consent
2. Willing to receive 13C-pyruvate DNP MRS and return for post-treatment evaluation for the scheduled follow up imaging about 1 week after initiation of chemotherapy.
3. Willing to receive therapy and follow-up as suggested by the tumor board and combined conference meeting in our institution
4. Presence of enlarged neck lymph nodes and/or spleen to serve as localized target for 3C-pyruvate DNP MRS

The exclusion criteria include:

1. Contraindicated to MRI study: such as cardiac pacemaker, cochlear implantation, metallic object within eyeball
2. Patients that refuse to, or has poor ability of understanding and comply study conditions, such as severe dementia or difficulty in mobility

The first stage planning Stage 1 started in the first year and is designed to evaluate the ability of 8 first-time diagnosed lymphoma patients referred from clinicians for 13C-pyruvate DNP MRS. The investigators expect to complete enrollment of the first 8 patients in the first year.

13C-Pyruvate DNP MRS scanning protocol for both Stage 1 and Stage 2: The MRI scanning protocol for both Stage 1 and Stage 2 are detailed as below Supplementary Appendix 1.

13C-Pyruvate DNP MRS Data Analysis and Post-processing : The MRI post-processing methods for both Stage 1 and Stage 2 are detailed as below Supplementary Appendix 2.

Expected completion of two stages For stage 1: The investigators expect to complete imaging for the 8 patients by the end of first year.

For Stage 2: The investigators expect to complete imaging for the 8 patients by the end of the second year.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide signed informed consent
2. Willing to receive 13C-pyruvate DNP MRS and return for post-treatment evaluation for the scheduled follow up imaging about 1 week after initiation of chemotherapy.
3. Willing to receive therapy and follow-up as suggested by the tumor board and combined conference meeting in our institution
4. Presence of enlarged neck lymph nodes and/or spleen to serve as localized target for 3C-pyruvate DNP MRS

The exclusion criteria include:

1. Contraindicated to MRI study: such as cardiac pacemaker, cochlear implantation, metallic object within eyeball
2. Patients that refuse to, or has poor ability of understanding and comply study conditions, such as severe dementia or difficulty in mobilit

Exclusion Criteria:

1. Contraindicated to MRI study: such as cardiac pacemaker, cochlear implantation, metallic object within eyeball
2. Patients that refuse to, or has poor ability of understanding and comply study conditions, such as severe dementia or difficulty in mobilit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of early treatment response of lymphoma patients using 13C pyruvate DNP MR spectroscopy | 2 years
  The changes in metabolic imaging biomarker levels
Assessment of early treatment response of lymphoma patients using 13C pyruvate DNP MR spectroscopy | 2 years
  The changes in metabolic tumor sizes

IPD SHARING:
Plan to Share IPD: Undecided